CLINICAL TRIAL: NCT05517382
Title: A Digital Game Targeting Suicide Prevention in Adolescents Who Report Substance Misuse (Formative Work and Pilot Study)
Brief Title: A Digital Game Targeting Suicide Prevention in Adolescents Who Report Substance Misuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000031180; 2KL2TR001862-06 (NIH)
Record Dates: First submitted 2022-08-23; First posted 2022-08-26 (Actual); Results first posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-03

CONDITIONS: Substance Misuse; Suicide
MeSH Terms: conditions — Suicide | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Eligible individuals will be assigned to either the 1) supportED group (n=30) or 2) control group (n=30).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supportED group (Experimental): Participants in this group will engage with the digital game for one session (~45min) and will receive NIDA and NIMH pamphlets on substance misuse and mental health for youth at the end of the session. Participants will use a dedicated device (e.g., tablet, laptop, or desktop) to access their digital experience on the web. The research staff and a school-based provider will be present to monitor gameplay, to provide support, if needed, and to field questions in person.
  Interventions: Other: supportED
- Control group (Other): Participants in this group will engage with a non-health-related game for one session (~45min) and will receive NIDA and NIMH pamphlets on substance misuse and mental health for youth at the end of the session. Participants will use a dedicated device (e.g., tablet, laptop, or desktop) to access their digital experience on the web. The research staff and a school-based provider will be present to monitor gameplay, to provide support, if needed, and to field questions in person.
  Interventions: Other: Control

INTERVENTIONS:
Other: supportED — suicide prevention videogame
  Arms: supportED group
Other: Control — non-health related videogame
  Arms: Control group

SUMMARY:
The primary aim of this study is to design and develop a digital game that models the process of a safety planning intervention. To do so, the investigators will explore and better understand peer or student perceptions around potential warning signs, coping strategies, and seeking help among youth who may be at greater risk of suicide due to misuse of substances. Focus groups/interviews with adolescents, young adults, adults, and school-based behavioral health providers will be conducted. Findings will inform the development of a digital intervention to reduce the risk of suicide among adolescents who misuse substances. Once a prototype of the game is developed, play-test focus groups with adolescents, college-aged youth, and school-based mental health providers will be conducted to finalize the intervention. Once finalized, the investigators will conduct a pilot study with 60 adolescents aged 13-19 to assess user experience, acceptability and feasibility of the digital game.

DETAILED DESCRIPTION:
Formative Work: In year 1, the aim is to design and develop a digital game that models the process of a safety planning intervention. To do so, the investigators will explore and better understand peer or student perceptions around potential warning signs, coping strategies, and seeking help among youth who may be at greater risk of suicide due to misuse of substances. Focus groups with adolescents, college-aged youth, and school-based mental health providers will be conducted. Findings will inform the development of a digital intervention to reduce the risk of suicide among adolescents who misuse substances. Once a prototype of the game is developed, the investigators will conduct play-test focus groups with adolescents and school-based mental health providers to finalize the digital game.

The focus of this clinical trial is the Pilot RCT: In year 2, the investigators will assess user experience, acceptability, and feasibility of the game as well as explore the following proximal outcomes such as but not limited to adolescent well-being, intentions to use a safety planning intervention, coping strategies, substance misuse in last 30 days, and associated risk factors related to suicidal risk (e.g., hopelessness, impulsivity, etc.).

ELIGIBILITY:
Inclusion Criteria:

* attend a high school that has a school-based behavioral health provider
* be fluent in reading English during the consent/assent process
* be willing to sit for a single session to complete pre-/post-assessments, engage with the game (~45min), and participate in a post-gameplay focus group (if in the experimental group) for 60min
* provide assent and parental/guardian consent (if<age 18).

Exclusion Criteria:

* Any student who is actively suicidal and/or moderately severe to severely depressed will be flagged and immediately connected to the school-based provider on site.
* If a student indicates moderately severe to severe symptoms of depression, student will be flagged and immediately connected to the school-based provider for a risk assessment and will follow appropriate school protocols. If student is cleared by the school-based provider, student may continue in the study and the school -based provider will follow up with student in two weeks.
* If a student screens positive for suicide (but is not acutely suicidal), student will be flagged and immediately connected to school-based provider for a risk assessment and will follow appropriate school protocols. If student is cleared by school-based provider, student may continue in study and the school-based provider will follow up with student in two weeks.
* If student is acutely suicidal, student will be flagged and immediately connected to school-based provider who will follow school protocol (e.g., contact 211, contact parent/guardian, etc.). They will be ineligible to participate in the study on this day. Student may not return to rescreen for participation for at least 2 weeks and only when they are no longer actively suicidal.

Rescreening: Participants will not have to repeat the questions related to static variables (such as demographics and past experiences), but the baseline assessment of dynamic variables will need to be repeated and meet eligibility requirements.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia-Santi F Fernandes, Ed.D., LPC, Principal Investigator — Yale University
Locations (1):
- Yale, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | supportED Group | Control Group
Started | 31 | 29
Completed Baseline Measures | 31 | 29
Completed 3 Month Follow up | 31 | 28
Completed | 31 | 28
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | supportED Group | Control Group | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.96 (1.02) | 16.63 (1.25) | 16.18 (1.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 14 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 19 | 41
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 1 | 1
  Race: Asian | 1 | 4 | 5
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Black or African American | 4 | 3 | 7
  Race: White | 17 | 12 | 29
  Race: More than one race | 4 | 4 | 8
  Race: Unknown or Not Reported | 4 | 5 | 9
  Race: Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Measuring Usability at Post-Gameplay
Description: Participants will complete surveys through a secured, data management system (RedCap). The Usefulness, Satisfaction, and Ease of Use Questionnaire (USE) is a validated, 30-item scale, where responses to system usability are measured on a scale from 1-7 where 1= strongly disagree and 7= strongly agree. Total score and subscales range 1-7. Higher scores indicate higher game usability.
Time Frame: Immediately after Gameplay, up to 30 minutes
Population: This outcome was not collected for the control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | supportED Group
Number analyzed (Participants) | 31
score on a scale
  Total score mean | 2.73 (0.52)
  Usefulness | 4.39 (1.70)
  Ease of use | 4.58 (1.50)
  Satisfaction | 4.69 (1.76)
  Ease of learning | 5.07 (1.76)

2. Primary Outcome: Assessing the Digital Experience at Post-Gameplay
Description: Participants were asked about negative and positive aspects of the digital experience. Data presented here are the count of overall positive and negative statements taken from an open ended question asking participants to provide up to 3 positive and 3 negative aspects of the digital experience.
Time Frame: Immediately after Gameplay, up to 30 minutes
Population: All coded statements provided in the open ended question. This outcome was not collected for the control arm.
Measure: Count of Units; unit: statements
Units Other Than Participants: statements
Arm/Group | supportED Group
Number analyzed (Participants) | 31
Number analyzed (statements) | 59
statements
  Positive | 32
  Negative | 27

3. Primary Outcome: Measuring User Experience at Post-Gameplay
Description: Participants will complete surveys through a secured data management system (RedCap). The User Engagement Scale-Short Form (UES-Short Form) is a validated, 12-item self report measure that assesses six domains of engagement where responses are measured on a 5-point likert scale where 1= strongly disagree and 5= strongly agree. Total score range 1-5.Higher scores indicate higher user engagement.
Time Frame: Immediately after Gameplay, up to 30 minutes
Population: This outcome was not collected for the control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | supportED Group
Number analyzed (Participants) | 31
score on a scale | 2.73 (0.52)

4. Primary Outcome: Measuring Acceptability at Post-Gameplay
Description: Participants will complete surveys through a secured data management system (RedCap). The Acceptability of Intervention Measure (AIM) is a validated, 4-item self-report measure of perceived acceptability where responses are measured on a 5-point likert scale where 1 = completely disagree and 5= completely agree. Higher scores indicate higher intervention acceptability. Note: This measure was removed from the final questionnaire due to redundancy.
Time Frame: Immediately after Gameplay, up to 30 minutes
Population: Survey was redundant and therefore removed. This data was not collected.
Arm/Group | supportED Group
Number analyzed (Participants) | 0

5. Primary Outcome: Measuring Feasibility at Post-Gameplay
Description: Feasibility will be measured through observation. Participants will also answer qualitative questions (e.g. does the intervention work? can the intervention be implemented in schools?) that will be developed by the study team. These questions are not a part of a larger scale. Minimal protocol deviations (Successful completion of protocols and procedures and minimal amendments through IRB) indicate feasibility of the digital game intervention. Data presented here are the number of deviations by type.
Time Frame: Immediately after Gameplay, up to 30 minutes
Measure: Number; unit: deviations
Arm/Group | supportED Group
Number analyzed (Participants) | 31
deviations
  RedCap Malfunction | 6
  Incomplete assent form signed off on | 2
  3-month form (first 3 measures) were completed at baseline. | 1

6. Secondary Outcome: Change From Baseline in Coping Strategies on Brief COPE Scale at Post-gameplay and 3-months
Description: Participants will complete surveys through a secured, data management system (RedCap). Brief Coping Orientation to Problems Experienced (Brief-COPE) adaptive and maladaptive subscales are validated, 28- item, 4-point self-report measures. Brief COPE measures assess 14 conceptually different coping reactions. Responses are measured on a 4-point likert scale where 1= I haven't been doing this at all and 4= I've been doing this a lot. Scores are summed to achieve total score with a range of 28-112. Higher scores indicate increased utilization of coping strategies within and across domains.
Time Frame: Baseline, Immediately after Gameplay (up to 30 minutes), and at 3-Months.
Population: one participant did not complete 3 month follow up
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | supportED Group | Control Group
Number analyzed (Participants) | 31 | 29
score on a scale
  Baseline | 60.72 [57.26 to 64.17] | 60.72 [57.26 to 64.17]
  Post gameplay | 58.92 [55.19 to 62.64] | 57.02 [53.25 to 60.79]
  3 months: number analyzed (Participants) | 31 | 28
  3 months | 63.36 [59.23 to 67.49] | 62.91 [58.48 to 67.34]

7. Secondary Outcome: Change From Baseline in Emotion Regulation at Post-gameplay and 3-months
Description: Participants will complete surveys through a secured, data management system (RedCap). State-Difficulties in Emotion Regulation (S-DERS) is a validated, 21-item self-report measure. Responses are measured on a 5-point likert scale where 1= almost never and 5= almost always. Scores are summed for total score range of 21-105. Higher scores suggest greater problems with emotion regulation.
Time Frame: Baseline, Immediately after Gameplay (up to 30 minutes), and at 3-months
Population: one participant did not complete 3 month follow up
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | supportED Group | Control Group
Number analyzed (Participants) | 31 | 29
score on a scale
  Baseline | 45.18 [42.34 to 48.02] | 45.18 [42.34 to 48.02]
  Post gameplay | 40.72 [37.95 to 43.50] | 42.84 [39.99 to 45.69]
  3 months: number analyzed (Participants) | 31 | 28
  3 months | 42.72 [39.35 to 46.10] | 45.58 [42.08 to 49.08]

8. Secondary Outcome: Percentage of Adolescents Thriving Post-gameplay and 3-months.
Description: Participants will complete surveys through a secured, data management system (RedCap). The Adolescent Well-Being assessment is a validated, 15-item school-based, self-report measure with 11-items focused on well being, and 5-items focused on student demographics. Higher scores indicate increased adolescent well-being. Data presented here is the difference in the change in the percentage of participants who were rated as "thriving" based on scores.
Time Frame: Immediately after Gameplay (up to 30 minutes), and at 3-Months.
Population: one participant did not complete 3 month follow up
Measure: Number; unit: percentage of participants
Arm/Group | supportED Group | Control Group
Number analyzed (Participants) | 31 | 29
percentage of participants
  Baseline | 41.9 | 58.6
  Post game | 51.6 | 58.6
  3 month: number analyzed (Participants) | 31 | 28
  3 month | 58.1 | 57.1
Statistical Analysis 1: Comparison: supportED Group vs Control Group; At baseline; Test type: Superiority; p = 0.20, t-test, 2 sided
Statistical Analysis 2: Comparison: supportED Group vs Control Group; At Post game; Test type: Superiority; p = 0.59, t-test, 2 sided
Statistical Analysis 3: Comparison: supportED Group vs Control Group; At 3 month; Test type: Superiority; p = 0.94, t-test, 2 sided
Statistical Analysis 4: Comparison: supportED Group vs Control Group; Test type: Superiority; p = 0.55, GEE; Controlling for baseline thriving status, this reflects the interaction between the intervention group and time

9. Secondary Outcome: Change From Baseline in Mindfulness at Post Gameplay and 3-months
Description: Participants will complete surveys through a secured, data management system (RedCap). The Five Facet Mindfulness Questionnaire (FFMQ) FFMQ is a validated, 15-item self-report measure that assesses facets of mindfulness. Responses are measured on a 5 point-likert scale where 1= never or very rarely true, and 5= very often or always true. Total score range 0-15. Higher scores indicate higher levels of mindfulness.
Time Frame: Baseline, Immediately after Gameplay (up to 30 minutes), and at 3-months
Population: one participant did not complete 3 month follow up
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | supportED Group | Control Group
Number analyzed (Participants) | 31 | 29
score on a scale
  Baseline | 3.47 [3.35 to 3.59] | 3.47 [3.35 to 3.59]
  Post gameplay | 3.46 [3.32 to 3.59] | 3.37 [3.23 to 3.50]
  3 months | 3.44 [3.29 to 3.59] | 3.28 [3.13 to 3.43]
Statistical Analysis 1: Comparison: supportED Group vs Control Group; At post game; Test type: Superiority; p = 0.1759, Mixed Models Analysis; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.23 to 0.04] — Group effect
Statistical Analysis 2: Comparison: supportED Group vs Control Group; At 3 month; Test type: Superiority; p = 0.0857, Mixed Models Analysis; Mean Difference (Net) = -0.16, 95% CI 2-sided [-0.35 to 0.02] — Group effect

10. Secondary Outcome: Change From Baseline in Intentions to Use a Safety Approach at Post-gameplay and 3-months.
Description: Participants will complete surveys through a secured, data management system (RedCap). Intentions to use a safety plan is a 7-item measure. Responses are measured on a 5-point likert scale where 1= strongly disagree and 5= strongly agree. Items are summed for a total score range of 7-35. Higher scores indicate increased intentions to use a safety planning approach.
Time Frame: Baseline, Immediately after Gameplay (up to 30 minutes), and at 3-Months.
Population: one participant did not complete 3 month follow up
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | supportED Group | Control Group
Number analyzed (Participants) | 31 | 29
score on a scale
  Baseline | 15.78 [14.33 to 17.24] | 15.78 [14.33 to 17.24]
  Post gameplay | 17.84 [16.12 to 19.55] | 16.38 [14.63 to 18.13]
  3 months: number analyzed (Participants) | 31 | 28
  3 months | 16.65 [13.99 to 19.31] | 17.59 [14.81 to 20.38]

11. Secondary Outcome: Change From Baseline in Knowledge About the Safety Planning Approach at Post-gameplay and 3-months.
Description: Participants will complete surveys through a secured, data management system (RedCap). 6-items will assess learning goals of the intervention developed by the study team (e.g. warning signs, coping strategies, resources for support). These items are not apart of a larger scale. Total score range 0-8. Higher scores indicate increased knowledge about gameplay content.
Time Frame: Baseline, Immediately after Gameplay (up to 30 minutes), and at 3-Months
Population: one participant did not complete 3 month follow up
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | supportED Group | Control Group
Number analyzed (Participants) | 31 | 29
score on a scale
  Baseline | 6.32 [5.92 to 6.71] | 6.32 [5.92 to 6.71]
  Post gameplay | 6.3 [5.78 to 6.82] | 6.23 [5.7 to 6.76]
  3 months: number analyzed (Participants) | 31 | 28
  3 months | 6.27 [5.74 to 6.81] | 6.13 [5.58 to 6.68]

12. Secondary Outcome: Change From Baseline in Severity of Suicidal Thoughts and Associative Behaviors on Concise Health Risk Tracking Self-Report (CHRT-SR) at 3-months.
Description: Participants will complete surveys through a secured, data management system (RedCap). Concise Health Risk Tracking Self-Report (CHRT-SR) is a validated, 14 item, 5-point self report measures comprised of the following subscales: Propensity, Impulsivity, and Suicidal Thoughts. Responses are measured on a 5-point likert scale where 0= strongly disagree and 4= strongly agree. Total score range of 0-56. Higher scores indicate increased severity of suicidal thoughts and associative behaviors.
Time Frame: Baseline, and at 3-Months.
Population: one participant did not complete 3 month follow up
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | supportED Group | Control Group
Number analyzed (Participants) | 31 | 29
score on a scale
  Baseline | 9.33 [7.23 to 11.43] | 9.33 [7.23 to 11.43]
  3 months: number analyzed (Participants) | 31 | 28
  3 months | 8.26 [5.61 to 10.91] | 7.24 [4.44 to 10.04]

13. Secondary Outcome: Change From Baseline in Anxiety at 3-months.
Description: Participants will complete surveys through a secured, data management system (RedCap). The General Anxiety Disorder-7 (GAD-7) is a validated, 7-item self report measure that assesses symptoms of anxiety. Responses are measured on a 4-point likert scale where 0=not at all and 3=nearly everyday. Item scores are summed with a total score ranging from 0 to 21: 0-4 Minimal anxiety; 5-9 Mild anxiety; 10-14 Moderate anxiety; 15-21 Severe anxiety. Higher scores indicate increased levels of anxiety.
Time Frame: Baseline, and at 3-Months.
Population: one participant did not complete 3 month follow up
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | supportED Group | Control Group
Number analyzed (Participants) | 31 | 29
score on a scale
  Baseline | 5.25 [3.84 to 6.66] | 5.25 [3.84 to 6.66]
  3 month: number analyzed (Participants) | 31 | 28
  3 month | 3.59 [2.10 to 5.08] | 4.41 [2.84 to 5.99]

14. Secondary Outcome: Change From Baseline in Depression at 3-months.
Description: Participants will complete surveys through a secured, data management system (RedCap). The Patient Health Questionnaire-9 (PHQ-9) is a validated, 9-item self report measure that assesses symptoms of depression. The total score on the PHQ-9 ranges from 0 to 27. Higher scores indicate increased levels of depression.
Time Frame: Baseline, and at 3-Months.
Population: one participant did not complete 3 month follow up
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | supportED Group | Control Group
Number analyzed (Participants) | 31 | 29
score on a scale
  Baseline | 5.25 [3.87 to 6.63] | 5.25 [3.87 to 6.63]
  3 month: number analyzed (Participants) | 31 | 28
  3 month | 3.96 [2.36 to 5.56] | 4.97 [3.29 to 6.65]

15. Secondary Outcome: Change From Baseline in Help-Seeking Behavior at Post-gameplay and 3-months.
Description: Participants will complete surveys through a secured, data management system (RedCap). The General Help Seeking Questionnaire (GHSQ) is a validated, 20-item self-report measure that assesses professional and non professional help seeking behaviors. Responses are measured on a 7-point likert scale where 1=extremely unlikely and 7=extremely likely. Total score range 20-140. Higher scores indicate increased help-seeking behavior.
Time Frame: Baseline, Immediately after Gameplay (up to 30 minutes), and at 3-Months.
Population: one participant did not complete 3 month follow up
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | supportED Group | Control Group
Number analyzed (Participants) | 31 | 29
score on a scale
  Baseline | 41.02 [38.16 to 43.87] | 41.02 [38.16 to 43.87]
  Post gameplay | 42.21 [39.2 to 45.22] | 42.53 [39.49 to 45.58]
  3 month: number analyzed (Participants) | 31 | 28
  3 month | 43.25 [39.79 to 46.71] | 42.57 [38.97 to 46.18]

16. Secondary Outcome: Mean Number of Days of Substance Misuse in the Past 30 Days
Description: Participants will complete surveys through a secured, data management system (RedCap). Substance misuse of alcohol, tobacco and marijuana in the past 30-days will be measured. These measures are self-reported. Responses indicate frequency of use within past 30-days.
Time Frame: Baseline, and at 3-Months.
Population: One participant did not complete 3 month follow up
Measure: Mean (Standard Deviation); unit: days
Arm/Group | supportED Group | Control Group
Number analyzed (Participants) | 31 | 29
days
  Baseline-Alcohol | 0.0322581 (0.1796053) | 0.137931 (0.5157614)
  3 months-Alcohol: number analyzed (Participants) | 31 | 28
  3 months-Alcohol | 0 (0) | 0 (0)
  Baseline-Tobacco | 0 (0) | 0 (0)
  3 month-Tobacco: number analyzed (Participants) | 31 | 28
  3 month-Tobacco | 0 (0) | 0 (0)
  Baseline-Marijuana | 0 (0) | 0 (0)
  3 month-Marijuana: number analyzed (Participants) | 31 | 28
  3 month-Marijuana | 0 (0) | 0 (0)

17. Other Pre Specified Outcome: Change From Baseline in Suicide Risk at 3-months
Description: The Ask Suicide Screen Questions (ASQ) is a validated 5-question screening tool to determine suicide risk.
Time Frame: Baseline, and at 3-Months.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 3 months
Arm/Group | supportED Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 0/31 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT05517382/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT05517382/ICF_001.pdf